CLINICAL TRIAL: NCT01870583
Title: Comparison of Surgical Skin Preps During Cesarean Deliveries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, David Garry, Co-Director Obstetrics & MFM service Wakefield Division, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CCI#12-07-248
Record Dates: First submitted 2013-06-03; First posted 2013-06-06 (Estimated); Results first posted 2017-06-19 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Surgical Site Infection Following Cesarean Delivery
Keywords: Cesarean delivery; Surgical site infection; Pregnancy; Postpartum
MeSH Terms: conditions — Surgical Wound Infection | interventions — Povidone-Iodine; Chlorhexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Combination iodine and chlorhexidine (Active Comparator): The combincation skin preparation will utilize the iodine based preparation first followed by the chlorhexidine based skin preparation prior to cesarean delivery.
  Interventions: Drug: Combination iodine and chlorhexidine
- Chlorhexidine (Active Comparator): Chlorhexidine based skin preparation solution applied to skin prior to cesarean delivery
  Interventions: Drug: Chlorhexidine
- Iodine povidone (Active Comparator): Iodine povidone based skin preparation solution applied to skin prior to cesarean delivery
  Interventions: Drug: Iodine povidone

INTERVENTIONS:
Drug: Iodine povidone — Iodine skin preparation solution prior to cesarean delivery
  Arms: Iodine povidone
Drug: Chlorhexidine — Chlorhexidine skin preparation solution prior to cesarean delivery
  Arms: Chlorhexidine
Drug: Combination iodine and chlorhexidine — Combination iodine povidone and chlorhexidine skin preparation solution prior to cesarean delivery
  Arms: Combination iodine and chlorhexidine

SUMMARY:
In women that undergo non-emergency cesarean delivery, we are comparing the skin preparation solutions for best outcome of surgical site infection. The three different solutions are: Group 1: Iodine povidone based skin preparation solution. Group 2: Chlorhexidine based skin preparation solution or Group 3: Combination usage of iodine povidone and chlorhexidine based skin preparation solutions. Women are prospectively randomized to one of the three groups and followed until thier postpartum visit at 6-8 weeks following delivery.

DETAILED DESCRIPTION:
Currently the skin preparation solutions currently in use for cesarean delivery are chlorhexidine-alcohol based solutions or iodine povidone solutions There had been no recommendations of which surgical skin prep wound be best utilized for cesarean delivery, especially if the patient has risk factors for surgical site infection. Chlorhexidine solution has been reported to take minimal of 2 minutes after application to decrease the bacterial load, and continue to decrease the bacteria load up to 1 hour. Iodine povidone solution has been reported to be completely effective within 4 minutes of application. Patient's risk factor for surgical site infection, including obesity, history of incision complications, maternal diabetes, chorioamnionitis, potentially influence which surgical skin prep to be applied. Finally, the majority of postpartum infections manifest after hospital discharge and most of these post-discharge infections are diagnosed and treated entirely in the ambulatory setting, without the patients' returning to the hospital.

The purpose of the study is:

1. To compare chlorhexidine based solution, iodine povidone solution, and combination of both agents in cesarean delivery skin preparation solution for prevention of surgical site infection (SSI)
2. To determine if surgical site infection (SSI) risk factors should guide selection of one specific surgical skin preparation solution.

This will be a prospective randomized observational study of the women presenting for care to the Montefiore Medical Center. All patients will undergo routine obstetrical care and preparation for cesarean delivery as if they were not participating in this research study. All patients in the study will receive the pre-operative intravenous antibiotics pre-operatively as part of departmental protocol for cesarean delivery.

The patients will be randomized after informed consent obtained into one of three groups: Group 1: Iodine povidone based skin preparation solution. Group 2: Chlorhexidine based skin preparation solution or Group 3: Combination usage of iodine povidone and chlorhexidine based skin preparation solutions. Sequentially numbered envelopes will contain the group of randomization for the patient created by a computer generated program which will occur prior to commencement of the study.

Surgical preparation will follow the departmental protocol as if the patient were not in the study with exception of the skin preparation. Once the patient is randomized to the skin preparation group, the corresponding skin preparation solution will be used in accordance to manufacturer's guidelines for the product and Departmental protocol. If randomized to group 3 (combination), the iodine based preparation will occur first followed by the chlorhexidine based skin preparation. All groups will wait a minimal of 4 minutes prior to skin incision after application of skin prep, and all patients will be surgically draped with the standard drapes as if not participating in a study. Cesarean delivery will occur following the technique of the surgeon, including skin closure method, suture or staples.

All patients will be followed until the routine postpartum visit occurs at 6-8 weeks following delivery. Postpartum visit information will be extracted from the medical record. If no postpartum visit occurs, the patient will be contacted by telephone at 8 weeks post delivery and asked about any incisional complications which may have occurred and required treatment by as physician or healthcare provider in the office or hospital.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age > 37 weeks 0/7 days
* Non-emergency indication for cesarean

Exclusion Criteria:

* Urogenital tract infection within 2 weeks prior to surgery
* Chronic oral or injectable steroid use (> 2 weeks)
* Emergency cesarean delivery
* Participation in another research study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1404 (Actual)
Dates: Start 2013-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Wallach, CIP, Study Chair — Einstein IRB
Locations (2):
- United States (2):
  - Montefiore Medical Center Weiler Division, The Bronx, New York
  - Montefiore Medical Center Wakefield Division, The Bronx, New York

REFERENCES:
- [Background] Zinn J, Jenkins JB, Harrelson B, Wrenn C, Haynes E, Small N. Differences in intraoperative prep solutions: a retrospective chart review. AORN J. 2013 May;97(5):552-8. doi: 10.1016/j.aorn.2013.03.006. PMID 23622828
- [Background] Berkelman RL, Holland BW, Anderson RL. Increased bactericidal activity of dilute preparations of povidone-iodine solutions. J Clin Microbiol. 1982 Apr;15(4):635-9. doi: 10.1128/jcm.15.4.635-639.1982. PMID 7040461
- [Background] Stinner DJ, Krueger CA, Masini BD, Wenke JC. Time-dependent effect of chlorhexidine surgical prep. J Hosp Infect. 2011 Dec;79(4):313-6. doi: 10.1016/j.jhin.2011.08.016. Epub 2011 Oct 15. PMID 22000737
- [Background] Olsen MA, Butler AM, Willers DM, Gross GA, Hamilton BH, Fraser VJ. Attributable costs of surgical site infection and endometritis after low transverse cesarean delivery. Infect Control Hosp Epidemiol. 2010 Mar;31(3):276-82. doi: 10.1086/650755. PMID 20102279
- [Background] Gong SP, Guo HX, Zhou HZ, Chen L, Yu YH. Morbidity and risk factors for surgical site infection following cesarean section in Guangdong Province, China. J Obstet Gynaecol Res. 2012 Mar;38(3):509-15. doi: 10.1111/j.1447-0756.2011.01746.x. Epub 2012 Feb 22. PMID 22353388
- [Background] Miner AL, Sands KE, Yokoe DS, Freedman J, Thompson K, Livingston JM, Platt R. Enhanced identification of postoperative infections among outpatients. Emerg Infect Dis. 2004 Nov;10(11):1931-7. doi: 10.3201/eid1011.040784. PMID 15550202
- [Background] Opoien HK, Valbo A, Grinde-Andersen A, Walberg M. Post-cesarean surgical site infections according to CDC standards: rates and risk factors. A prospective cohort study. Acta Obstet Gynecol Scand. 2007;86(9):1097-102. doi: 10.1080/00016340701515225. PMID 17712651
- [Background] Lobdell KW, Stamou S, Sanchez JA. Hospital-acquired infections. Surg Clin North Am. 2012 Feb;92(1):65-77. doi: 10.1016/j.suc.2011.11.003. Epub 2011 Dec 5. PMID 22269261
- [Background] Segal CG, Anderson JJ. Preoperative skin preparation of cardiac patients. AORN J. 2002 Nov;76(5):821-8. doi: 10.1016/s0001-2092(06)61035-1. PMID 12463081
- [Derived] Hadiati DR, Hakimi M, Nurdiati DS, Masuzawa Y, da Silva Lopes K, Ota E. Skin preparation for preventing infection following caesarean section. Cochrane Database Syst Rev. 2020 Jun 25;6(6):CD007462. doi: 10.1002/14651858.CD007462.pub5. PMID 32580252
- [Derived] Ngai IM, Van Arsdale A, Govindappagari S, Judge NE, Neto NK, Bernstein J, Bernstein PS, Garry DJ. Skin Preparation for Prevention of Surgical Site Infection After Cesarean Delivery: A Randomized Controlled Trial. Obstet Gynecol. 2015 Dec;126(6):1251-1257. doi: 10.1097/AOG.0000000000001118. PMID 26551196

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Combination Iodine and Chlorhexidine | Chlorhexidine | Iodine Povidone
Started | 467 | 474 | 463
Completed | 456 | 456 | 455
Not Completed | 11 | 18 | 8
Not completed — Protocol Violation | 0 | 5 | 3
Not completed — Lost to Follow-up | 11 | 13 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination Iodine and Chlorhexidine | Chlorhexidine | Iodine Povidone | Total
Number analyzed (Participants) | 467 | 474 | 463 | 1404
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.1 (5.9) | 30.3 (5.7) | 29.9 (6.0) | 30.2 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 467 | 474 | 463 | 1404
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 467 | 474 | 463 | 1404

OUTCOME MEASURES:

1. Primary Outcome: Cesarean Surgical Site Infection
Description: Surgical site infection will follow CDC guidelines: A) Superficial incisional surgical site infection B) Deep incisional surgical site infection or C) Organ/space surgical site infection.
Time Frame: 42 days after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Iodine and Chlorhexidine | Chlorhexidine | Iodine Povidone
Number analyzed (Participants) | 467 | 474 | 463
Participants
  Any SSI: Total combined | 18 | 21 | 21
  SSI: Superficial | 15 | 15 | 16
  SSI: Deep | 1 | 3 | 3
  SSI: Organ | 2 | 3 | 2

ADVERSE EVENTS:
Arm/Group | Combination Iodine and Chlorhexidine | Chlorhexidine | Iodine Povidone
All-Cause Mortality (participants affected / at risk) | 0/467 | 0/474 | 0/463
Serious Adverse Events (participants affected / at risk) | 2/467 | 3/474 | 2/463
Other Adverse Events (participants affected / at risk) | 0/467 | 0/474 | 0/463
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Iodine and Chlorhexidine (N=467) | Chlorhexidine (N=474) | Iodine Povidone (N=463)
Surgical site infection: organ (Infections and infestations) | 2 | 3 | 2 — Admissions to hospital for IV antibiotics. No relationship to skin preparation solution

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No